CLINICAL TRIAL: NCT04505631
Title: Follow-up of Respiratory Sequelae of Patients Hospitalized With SARS-CoV-2: a Prospective Multicenter Observational Study
Brief Title: Follow-up of Respiratory Sequelae of Hospitalized Patients With COVID-19
Acronym: SISCOVID
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Other Study IDs: GHRMSA 1052; IDRCB 2020-A01089-30 (Other: ANSM)
Record Dates: First submitted 2020-08-03; First posted 2020-08-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Covid19; Dyspnea
Keywords: COVID19; PNEUMOPATHY; DYSPNEA
MeSH Terms: conditions — COVID-19; Dyspnea; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this multicenter observational study is to describe respiratory sequelae of COVID-19 patients hospitalized for severe pneumonia requiring oxygen supply.

DETAILED DESCRIPTION:
Main objective To assess respiratory sequelae after SARS-CoV-2 infection in hospitalized patients with severe pneumonia requiring oxygen supply and followed up for 6 months after hospital discharge (see primary and secondary outcomes).

Secondary objectives

To describe pulmonary sequelae according to :

* the unit in which the patient was hospitalized,
* the maximum oxygen flow rate required during hospitalization,
* McCabe score,
* age,
* tobacco consumption,
* biological data (e.g. blood count, CRP, fibrinogen, LDH, albumin, D-dimer, ferritin),
* number of days from onset of symptoms to hospitalization,
* co-morbidities (e.g. diabetes, hypertension, coronary artery disease/heart failure, mild to moderate COPD/respiratory failure, overweight),
* concomitant treatments (e.g. non-steroidal anti-inflammatory drugs, corticosteroids, immunosuppressants, ACE inhibitors)
* specific drug treatments administered to treat COVID-19 infection,
* non-drug treatments (invasive ventilation, non-invasive ventilation, postural treatment) to manage respiratory disorders of COVID-19 infection.

To assess the impact of factors of social inequality on the severity of COVID-19 infection.

Conduct of research Patients who have been hospitalized for severe pneumonia due to CoV-2 SARS infection will be seen in consultation at approximately 3 and 6 months after hospital discharge, as per standard practice.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years old
* SARS-CoV-2 infection proven by RT-PCR and/or retrospective serology and/or a COVID-19 syndrome with evocative chest CT scan
* Hospitalized for severe pneumonia due to SARS-CoV-2 infection requiring oxygen supply

Exclusion criteria:

* Not hospitalized for a severe COVID-19 infection
* Absence of respiratory symptoms at V1 (3 months after hospital discharge), defined as: absence of residual exertional dyspnea and persistent pulmonary infiltrates on follow-up chest radiography at 1 month (if available), transcutaneous oxyhemoglobin saturation >94% and normal pulmonary auscultation
* Patient with pre-existing chronic lung disease prior to the first episode of COVID-19: chronic obstructive pulmonary disease confirmed by respiratory function testing with a forced expiratory volume in one second (FEV1) < 50% and/or a diffusing capacity for carbon monoxide (DLCO) < 60%, fibrotic lung disease or chronic respiratory failure (on long-term oxygen therapy)
* Opposition to participation in the study
* Patient under legal protection
* Patient not affiliated to/beneficiary of a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been hospitalized for severe pneumonia due to SARS-CoV-2 infection will be seen in consultation at approximately 3 and 6 months after hospital discharge, as per standard practice.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Presence of respiratory sequelae | 6 months after hospital discharge
  The presence of respiratory sequelae will be assessed by low dose thoracic tomodensitometry

SECONDARY OUTCOMES:
Presence of respiratory sequelae on low dose thoracic tomodensitometry | 3 months after hospital discharge
Forced vital capacity (FVC, %) | 6 months after hospital discharge
  Respiratory functional exploration
Forced vital capacity (FVC, %) | 3 months after hospital discharge
  Respiratory functional exploration
Forced expiratory volume in 1 second (FEV1, %) | 6 months after hospital discharge
  Respiratory functional exploration
Forced expiratory volume in 1 second (FEV1, %) | 3 months after hospital discharge
  Respiratory functional exploration
Tiffeneau-Pinelli index (FEV1/FVC, %) | 6 months after hospital discharge
  Respiratory functional exploration
Tiffeneau-Pinelli index (FEV1/FVC, %) | 3 months after hospital discharge
  Respiratory functional exploration
Total lung capacity (TLC, %) | 6 months after hospital discharge
  Respiratory functional exploration
Total lung capacity (TLC, %) | 3 months after hospital discharge
  Respiratory functional exploration
Residual volume (RV, %) | 6 months after hospital discharge
  Respiratory functional exploration
Residual volume (RV, %) | 3 months after hospital discharge
  Respiratory functional exploration
RV/TLC ratio (%) | 6 months after hospital discharge
  Respiratory functional exploration
RV/TLC ratio (%) | 3 months after hospital discharge
  Respiratory functional exploration
Maximal inspiratory pressure (MIP, %) | 6 months after hospital discharge
  Respiratory functional exploration
Maximal inspiratory pressure (MIP, %) | 3 months after hospital discharge
  Respiratory functional exploration
Maximal expiratory pressure (MEP, %) | 6 months after hospital discharge
  Respiratory functional exploration
Maximal expiratory pressure (MEP, %) | 3 months after hospital discharge
  Respiratory functional exploration
Diffusion capacity of the lungs for carbon monoxide (DLCO, %) | 6 months after hospital discharge
  Respiratory functional exploration
Diffusion capacity of the lungs for carbon monoxide (DLCO, %) | 3 months after hospital discharge
  Respiratory functional exploration
pH | 6 months after hospital discharge
  Arterial gasometry will be performed under ambient air and under oxygen
pH | 3 months after hospital discharge
  Arterial gasometry will be performed under ambient air and under oxygen
Arterial oxygen partial pressure (PaO2, mmHg) | 6 months after hospital discharge
  Arterial gasometry will be performed under ambient air and under oxygen
Arterial oxygen partial pressure (PaO2, mmHg) | 3 months after hospital discharge
  Arterial gasometry will be performed under ambient air and under oxygen
Arterial carbon dioxide partial pressure (PaCO2, mmHg) | 6 months after hospital discharge
  Arterial gasometry will be performed under ambient air and under oxygen
Arterial carbon dioxide partial pressure (PaCO2, mmHg) | 3 months after hospital discharge
  Arterial gasometry will be performed under ambient air and under oxygen
Bicarbonate concentration (mmol/L) | 6 months after hospital discharge
  Arterial gasometry will be performed under ambient air and under oxygen
Bicarbonate concentration (mmol/L) | 3 months after hospital discharge
  Arterial gasometry will be performed under ambient air and under oxygen
Arterial oxygen saturation (SaO2, %) | 6 months after hospital discharge
  Arterial gasometry will be performed under ambient air and under oxygen
Arterial oxygen saturation (SaO2, %) | 3 months after hospital discharge
  Arterial gasometry will be performed under ambient air and under oxygen
Six-minute walk test | 6 months after hospital discharge
  Six-minute walk test will be performed under ambient air and under oxygen
Six-minute walk test | 3 months after hospital discharge
  Six-minute walk test will be performed under ambient air and under oxygen

CONTACTS AND LOCATIONS:
Overall Officials: George-Daniel Calcaianu, MD, Principal Investigator — GHRMSA hospital
Locations (14):
- France (14):
  - Groupe Hospitalier de Mulhouse et de la Région Sud-Alsace, Mulhouse, Alsace
  - Centre Hospitalier de la Côte Basque - Bayonne, Bayonne
  - Centre Hospitalier Métropole Savoie, Chambéry
  - Centre Hospitalier Colmar, Colmar
  - Centre Hospitalier Douai, Douai
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Centre Hospitalier Départemental Vendée - La Roche sur Yon, La Roche-sur-Yon
  - Centre Hospitalier du Mans, Le Mans
  - Centre Hospitalier Robert Boulin - Libourne, Libourne
  - Centre Hospitalier Régional Metz-Thioville, Metz
  - Centre Hospitalier Annecy Genevois, Metz-Tessy
  - Centre Hospitalier Le Raincy Montfermeil, Montfermeil
  - Centre Hospitalier Régional Orléans, Orléans
  - Centre Hospitalier de Soissons, Soissons

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Calcaianu G, Degoul S, Michau B, Payen T, Gschwend A, Fore M, Iamandi C, Morel H, Oster JP, Bizieux A, Nocent-Ejnaini C, Carvallo C, Romanet S, Goupil F, Leurs A, Legrand MG, Portel L, Claustre J, Calcaianu M, Bresson D, Debieuvre D. Mid-term pulmonary sequelae after hospitalisation for COVID-19: The French SISCOVID cohort. Respir Med Res. 2022 Nov;82:100933. doi: 10.1016/j.resmer.2022.100933. Epub 2022 Jun 14. PMID 35905553